CLINICAL TRIAL: NCT02482857
Title: Optimal Dose of Acetylsalicylic Acid After Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASA-dos
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Bypass Surgery; Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acetylsalicylic acid 75 mg twice daily (Experimental): Aspirin 75 mg BID is a new experimental dosing regimen which has shown improved efficiency regarding laboratory parameters in several studies, mainly in diabetic patients.
  Interventions: Drug: Acetylsalicylic acid
- Acetylsalicylic acid 160 mg once daily (Active Comparator): Aspirin 160 mg OD is an accepted and used dosage after CABG.
  Interventions: Drug: Acetylsalicylic acid
- Acetylsalicylic acid 75 mg once daily (Active Comparator): Aspirin 75 mg OD is an accepted and used dosage after CABG.
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid — To compare BID dosing with OD dosing with clinically used aspirin dosages.
  Other Names: Aspirin

SUMMARY:
This is a single-center, open-label, randomized controlled trial. Patients with stable angina pectoris without use of dual antiplatelet therapy or anticoagulation therapy scheduled for coronary artery bypass grafting (CABG) at Karolinska University Hospital in Stockholm, Sweden will be eligible.

This study investigates in patients having undergone CABG whether increasing the dose or the frequency of acetylsalicylic acid (ASA) treatment improves the efficacy of ASA regarding platelet inhibition compared to the standard dosing for cardiovascular prevention (75 mg once daily) in the first three months after surgery. Patients will be randomly assigned to postoperative ASA dose 75mg once daily, 75mg twice daily or 160 mg once daily. The study dose ASA will be started at hospital discharge and continued of three months. Blood samples for serum thromboxane B2 (TxB2) and other analyses will be taken before surgery, before discharge, and after one and three months. All available data will be collected prospectively. Informed consent will be obtained from patients meeting the inclusion criteria before the initiation of any study-specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease
* ≥18 years of age
* Scheduled to undergo elective CABG surgery
* Willing to participate and able to provide informed consent

Exclusion Criteria:

* Intake of drugs other than ASA that are known to influence platelet function, including nonsteroidal anti-inflammatory drugs (NSAIDs, including COX-2 selective anti-inflammatory drugs), GPIIbIIIa inhibitors, clopidogrel, dipyridamole, warfarin or acenocoumarol within 7 days of enrolment
* Hemorrhagic diathesis or known platelet dysfunction
* Chronic renal failure requiring dialysis
* Platelet count outside the 100 000 to 450 000/μL range
* Haemoglobin < 8g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Serum thromboxane B2 | 3 months

SECONDARY OUTCOMES:
Multiple electrode aggregometry platelet aggregation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hjemdahl, Professor, Principal Investigator — Karolinska University Hospital